CLINICAL TRIAL: NCT05973630
Title: A Phase 1-2, Open-label Study to Evaluate the Safety of Intravenous ATA-200, an Adeno-associated Viral Vector Carrying the Human SGCG Gene, in Patients With Gamma-sarcoglycanopathy (LGMDR5)
Brief Title: ATA-200 Gene Therapy Trial in Patients With LGMDR5
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atamyo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATA-003-GSAR
Record Dates: First submitted 2023-07-24; First posted 2023-08-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: LGMD2C
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): ATA-200 Dose : 1.0E+14 vg/Kg, solution for injection, single IV infusion over 2h
  Interventions: Biological: ATA-200

INTERVENTIONS:
Biological: ATA-200 — single intravenous infusion

SUMMARY:
The purpose of ATA-003-GSAR study is to evaluate the safety and tolerability of a single intravenous infusion of ATA-200 in pediatric patients with limb girdle muscular dystrophy type 2c/R5 (LGMD R5).

DETAILED DESCRIPTION:
This is a multicenter Phase 1b assessing the safety and tolerability of intravenous ATA-200 for the treatment of LGMDR5.

The study will enroll ambulant patients with LGMDR5. Patients will be enrolled sequentially and enrollment will be staggered with at least 4-week interval between 2 patient treatments. Patients will receive a potentially effective dose corresponding to the minimum effective dose (MED) in preclinical studies.

Time point of primary interest for safety evaluation and dose selection for future studies is at 6 months.

All subjects will be followed up for an additional 4.5 years after completion of the initial evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of LGMDR5 before age of 10, based on clinical presentation and genotyping
* Ambulant male or female patients aged 6 to less than 12 years of age at screening
* Able to perform the 10-meter walk test (10MWT) in less than 15 sec and to rise from chair with or without arm support

Exclusion Criteria:

* Detectable neutralizing antibodies against AAV8
* Cardiomyopathy with left ventricular ejection fraction (LVEF) < 50%
* Respiratory assistance
* Concomitant medical condition that might interfere with LGMDR5 evolution
* Acute illness within 4 weeks of anticipated IMP administration
* Current participation in another clinical trial with investigational medicinal product
* Previous participation in gene and cell therapy trials
* Any condition that would contraindicate immunosuppressant treatment
* Presence of any permanent items (e.g., metal braces) precluding undergoing MRI
* Any vaccination 1 month prior to planned IMP administration
* Serology consistent with HIV exposure or active hepatitis B or C infection
* Grade 2 or higher lab abnormalities for liver function tests, creatinine, hemogram and coagulation

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 0-6 months
  Collection of adverse events at each visit
Incidence of treatment-emergent adverse events, | 0-6 months
  Collection of adverse events at each visit
Incidence of serious adverse events | 0-6 months
  Collection of adverse events at each visits

CONTACTS AND LOCATIONS:
Locations (1):
- Child Health Research Institute, Gainsville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided